CLINICAL TRIAL: NCT00309101
Title: FK506 Phase 3 Study: An Open Study for Steroid Resistant, Non-Thymectomized MG Patients
Brief Title: An Open Study for Steroid Resistant, Non-Thymectomized MG Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F506-CL-0602
Record Dates: First submitted 2006-03-29; First posted 2006-03-31 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Myasthenia Gravis
Keywords: Tacrolimus; Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Tacrolimus

ARMS (1):
- 1. tacrolimus (Experimental)
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: tacrolimus — Oral
  Other Names: FK506; Prograf

SUMMARY:
The purpose of the study is to investigate the efficacy and safety for steroid resistant, non-thymectomized MG patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as myasthenia gravis
* Those whose MG symptoms are not controlled by the treatment with prednisone

Exclusion Criteria:

* Those who had undergone thymectomy

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2006-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Improvement of clinical symptoms | 28 Weeks

SECONDARY OUTCOMES:
Improvement of daily activity | 28 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (9):
- Japan (9):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Hokuriku Region
  - Kansai Region
  - Kanto Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region